CLINICAL TRIAL: NCT01598090
Title: A Phase 3 Blinded Randomized Study of Peginterferon Lambda-1a and Ribavirin Compared to Peginterferon Alfa-2a and Ribavirin, Each Administered With Telaprevir in Subjects With Genotype-1 Chronic Hepatitis C Who Are Treatment-naive or Relapsed on Prior Treatment With Peginterferon Alfa-2a and Ribavirin
Brief Title: Phase 3 Efficacy and Safety Study of Peginterferon Lambda-1a and Ribavirin With Telaprevir
Acronym: PEDESTAL
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AI452-020; 2011-004695-11 (EudraCT Number)
Record Dates: First submitted 2012-05-09; First posted 2012-05-15 (Estimated); Results first posted 2019-05-21 (Actual); Last update posted 2019-07-31 (Actual); Status verified 2019-07

CONDITIONS: Hepatitis C Virus
MeSH Terms: conditions — Hepatitis C | interventions — peginterferon lambda-1a; peginterferon alfa-2a; Ribavirin; telaprevir

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Part A: Peginterferon Lambda-1a + RBV + TVR (Experimental)
  Interventions: Biological: Peginterferon Lambda-1a; Drug: Ribavirin; Drug: Telaprevir
- Part B (Arm 1): Peginterferon Lambda-1a + RBV + TVR (Experimental)
  Interventions: Biological: Peginterferon Lambda-1a; Drug: Ribavirin; Drug: Telaprevir
- Part B (Arm 2): Peginterferon Lambda-2a + RBV + TVR (Experimental)
  Interventions: Biological: Peginterferon Alfa-2a; Drug: Ribavirin; Drug: Telaprevir

INTERVENTIONS:
Biological: Peginterferon Lambda-1a — Syringes, subcutaneous (SC), 180μg, Once weekly, 24 or 48 weeks depending on response
  Arms: Part A: Peginterferon Lambda-1a + RBV + TVR; Part B (Arm 1): Peginterferon Lambda-1a + RBV + TVR
Biological: Peginterferon Alfa-2a — Syringes, SC, 180μg, Once weekly, 24 or 48 weeks depending on response
  Other Names: Pegasys
  Arms: Part B (Arm 2): Peginterferon Lambda-2a + RBV + TVR
Drug: Ribavirin — Tablets, Oral, 1000 or 1200 mg based on weight, twice daily, 24 or 48 weeks depending on response
Drug: Telaprevir — Tablets, Oral, 750 mg, three times a day, 12 weeks only
  Other Names: Incivek

SUMMARY:
The purpose of this study is to determine whether Peginterferon Lambda-1a (Lambda) combined with Ribavirin (RBV) and Telaprevir (TVR) is effective in the treatment of chronic Hepatitis C (CHC) compared to Peginterferon Alfa-2a (alfa-2a) combined with RBV and Telaprevir.

ELIGIBILITY:
For more information regarding BMS clinical trial participation, please visit www.BMSStudyConnect.com.

Inclusion Criteria:

* Chronic hepatitis C genotype 1. GT-1b Capped at 50 % of naïve subjects
* Naives to prior anti-HCV therapy [Interferon (IFN) and direct antiviral agent (DAA) based]
* Relapsers (defined as subjects who had undetectable HCV ribonucleic acid (RNA) on prior treatment regimen of alfa-2a/RBV and Hepatitis C Virus (HCV) RNA > 25IU/mL after discontinuation of treatment). Capped at 20%
* HCV RNA ≥ 100,000 IU/mL
* Subjects with compensated cirrhosis can be enrolled and will be capped at approximately 10%
* Seronegative for human immunodeficiency virus (HIV) and hepatitis B surface antigen (HBsAg)
* Men or women, 18-70 years of age

Exclusion Criteria:

* Chronic liver disease due to causes other than chronic HCV
* Current or past evidence of decompensation
* Conditions that preclude the use of Alfa/RBV/TVR per respective labels
* Diagnosed or suspected hepatocellular carcinoma

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 881 (Actual)
Dates: Start 2012-06-14 (Actual); Primary Completion 2015-02-04 (Actual); Study Completion 2015-05-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (88):
- United States (28):
  - Birmingham Gastroenterology Associates, P.C., Birmingham, Alabama
  - The Kirklin Clinic, Birmingham, Alabama
  - The University Of Alabama Of Birmingham, Birmingham, Alabama
  - Anaheim Clinical Trials Llc, Anaheim, California
  - Sc Clinical Research, Inc., Garden Grove, California
  - Va Long Beach Healthcare System, Long Beach, California
  - Cedars Sinai Medical Center, Los Angeles, California
  - Va Greater Los Angeles Healthcare System, Los Angeles, California
  - University Of California, San Francisco/Sf General Hospital, San Francisco, California
  - South Bay Ge Medical Group, Torrance, California
  - Orlando Va Medical Center, Orlando, Florida
  - Orlando Clinical Research Center, Orlando, Florida
  - Infectious Disease Research Institute, Inc., Tampa, Florida
  - Gastrointestinal Specialists Of Georgia Pc, Marietta, Georgia
  - Mercy Medical Center, Baltimore, Maryland
  - Saint Luke'S Transplant Specialists, Kansas City, Missouri
  - Saint Louis University, St Louis, Missouri
  - Carolinas Medical Center, Charlotte, North Carolina
  - Options Health Research, Llc, Tulsa, Oklahoma
  - Healthcare Research Consultants, Tulsa, Oklahoma
  - Gastro One, Germantown, Tennessee
  - Texas Clinical Research Institute, Arlington, Texas
  - Brooke Army Medical Center, Fort Sam Houston, Texas
  - Alamo Medical Research, San Antonio, Texas
  - Clinical Research Centers Of America, Murray, Utah
  - Metropolitan Research, Annandale, Virginia
  - Bon Secours St. Mary'S Hospital Of Richmond, Inc., Newport News, Virginia
  - Digestive And Liver Disease Specialists, Norfolk, Virginia
- Austria (2):
  - Local Institution, Graz
  - Local Institution, Linz
- Belgium (4):
  - Local Institution, Brussels
  - Local Institution, Edegem
  - Local Institution, Leuven
  - Local Institution, Liège
- Brazil (6):
  - Local Institution, Salvador, Estado de Bahia
  - Local Institution, Curitiba, Paraná
  - Local Institution, Porto Alegre, Rio Grande do Sul
  - Local Institution, Botucatu, São Paulo
  - Local Institution, Rio de Janeiro
  - Local Institution, São Paulo
- Canada (6):
  - University Of Calgary, Calgary, Alberta
  - Liver And Intestinal Research Centre (Lair), Vancouver, British Columbia
  - Gastrointestinal Research Institute (G.I.R.I.), Vancouver, British Columbia
  - Percuro Clinical Research Ltd, Victoria, British Columbia
  - Toronto General Hospital, Toronto, Ontario
  - Hopital Maisonneuve-Rosemont, Montreal, Quebec
- Czechia (2):
  - Local Institution, Hradec Králové
  - Local Institution, Prague
- France (6):
  - Local Institution, Orléans
  - Local Institution, Poitiers
  - Local Institution, Rennes
  - Local Institution, Rouen
  - Local Institution, Toulouse
  - Local Institution, Villejuif
- Germany (7):
  - Local Institution, Berlin
  - Local Institution, Essen
  - Local Institution, Frankfurt
  - Local Institution, Hamburg
  - Local Institution, Hanover
  - Local Institution, Münster
  - Local Institution, Ulm
- Israel (4):
  - Local Institution, Haifa
  - Local Institution, Jerusalem
  - Local Institution, Nazareth
  - Local Institution, Ramat Gan
- Italy (5):
  - Local Institution, Bergamo
  - Local Institution, Cisanello (pisa)
  - Local Institution, Milan
  - Local Institution, Roma
  - Local Institution, Torino
- Poland (6):
  - Local Institution, Bialystok
  - Local Institution, Kielce
  - Local Institution, Mysłowice
  - Local Institution, Racibórz
  - Local Institution, Wroclaw
  - Local Institution, Łańcut
- Russia (4):
  - Local Institution, Kazan', Tatarstan Republic
  - Local Institution, Moscow
  - Local Institution, Saint Petersburg
  - Local Institution, Stavropol
- Spain (5):
  - Local Institution, A Coruña
  - Local Institution, Alicante
  - Local Institution, Donostia / San Sebastian
  - Local Institution, Santiago de Compostela
  - Local Institution, Seville
- Switzerland (2):
  - Local Institution, Basel
  - Local Institution, Zurich
- Local Institution, Birmingham, WEST Midlands, United Kingdom

REFERENCES:
- [Derived] Heim MH. 25 years of interferon-based treatment of chronic hepatitis C: an epoch coming to an end. Nat Rev Immunol. 2013 Jul;13(7):535-42. doi: 10.1038/nri3463. Epub 2013 Jun 7. PMID 23743475
- See also: BMS clinical trial educational resource — http://www.bms.com/studyconnect/Pages/home.aspx
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx
- See also: BMS Clinical Trial Patient Recruiting — http://bms.com/studyconnect/Pages/home.aspx

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Out of 881 participants who were enrolled, 648 were randomized and only 644 were treated. 27 participants were treated in Part A and 617 participants were treated in Part B of the study.
Groups:
- Part A: Peginterferon Lambda-1a + RBV + TVR (Open Label): Participants with genotype (GT) -1 chronic Hepatitis C virus infection received Peginterferon Lambda-1a 180 mcg subcutaneously, once weekly for 24 or 48 weeks depending on the extended rapid virologic response (eRVR); Ribavirin 1000 or 1200 mg (based on weight) tablets, orally daily in 2 divided doses for 24 or 48 weeks depending on the eRVR response; Telaprevir 750 mg tablets, orally three times a day for 12 weeks. Participants were followed-up for 48 weeks after treatment period.
- Part B: Peginterferon Lambda-1a + RBV + TVR: Participants who were either treatment naive or who were relapsers to previous Peginterferon alfa- 2a/ribavirin treatment received Peginterferon Lambda-1a 180 mcg subcutaneously, once weekly for 24 or 48 weeks depending on the extended rapid virologic response (eRVR); Ribavirin 1000 or 1200 mg (based on weight) tablets, orally daily in 2 divided doses for 24 or 48 weeks depending on the eRVR response; Telaprevir 750 mg tablets, orally three times a day for 12 weeks. Participants were followed-up for 48 weeks after treatment period.
- Part B: Peginterferon Alfa-2a + RBV + TVR: Participants who were either treatment naive or who were relapsers to previous Peginterferon alfa- 2a/ribavirin treatment received Peginterferon alfa-2a 180 mcg subcutaneously, once weekly for 24 or 48 weeks depending on the extended rapid virologic response (eRVR); Ribavirin 1000 or 1200 mg (based on weight) tablets, orally daily in 2 divided doses for 24 or 48 weeks depending on the eRVR response; Telaprevir 750 mg tablets, orally three times a day for 12 weeks. Participants were followed-up for 48 weeks after treatment period.
Period: Treatment Period
Arm/Group | Part A: Peginterferon Lambda-1a + RBV + TVR (Open Label) | Part B: Peginterferon Lambda-1a + RBV + TVR | Part B: Peginterferon Alfa-2a + RBV + TVR
Started | 27 | 411 | 206
Completed | 16 | 339 | 171
Not Completed | 11 | 72 | 35
Not completed — Poor/non-compliance | 0 | 2 | 0
Not completed — No longer meet study criteria | 0 | 1 | 0
Not completed — Lack of Efficacy | 5 | 14 | 6
Not completed — Adverse Event | 2 | 33 | 17
Not completed — Other reasons | 0 | 4 | 1
Not completed — Withdrawal by Subject | 3 | 13 | 10
Not completed — Lost to Follow-up | 1 | 5 | 1
Period: Follow-up Period
Arm/Group | Part A: Peginterferon Lambda-1a + RBV + TVR (Open Label) | Part B: Peginterferon Lambda-1a + RBV + TVR | Part B: Peginterferon Alfa-2a + RBV + TVR
Started | 26 (Includes 10 participants who re-joined from treatment period to follow-up period.) | 399 (Includes 60 participants who re-joined from treatment period to follow-up period.) | 199 (Includes 28 participants who re-joined from treatment period to follow-up period.)
Completed | 21 | 364 | 171
Not Completed | 5 | 35 | 28
Not completed — Death | 0 | 1 | 0
Not completed — No longer required per protocol | 1 | 3 | 2
Not completed — Not reported | 0 | 10 | 4
Not completed — Withdrawal by Subject | 0 | 3 | 2
Not completed — Other reasons | 2 | 8 | 8
Not completed — Lost to Follow-up | 2 | 10 | 12

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Part A: Peginterferon Lambda-1a + RBV + TVR (Open Label) | Part B: Peginterferon Lambda-1a + RBV + TVR | Part B: Peginterferon Alfa-2a + RBV + TVR | Total
Number analyzed (Participants) | 27 | 411 | 206 | 644
Age, Customized [Count of Participants; unit: Participants]
  <21 years | 0 | 5 | 2 | 7
  21 - <65 years | 27 | 392 | 197 | 616
  >=65 years | 0 | 14 | 7 | 21
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 152 | 80 | 241
  Male | 18 | 259 | 126 | 403

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Extended Rapid Virologic Response (eRVR) - Part A
Description: eRVR was defined as Hepatitis C virus (HCV) RNA level below the lower limit of quantitation, target not detected at Weeks 4 and 12 of treatment. HCV RNA level was measured using the Roche COBAS® TaqMan HCV Test v.2.0 (lower limit of quantitation =25 IU/mL; limit of detection ~ 10 IU/mL).
Time Frame: Assessed at Week 4 and Week 12, week 12 reported
Population: The analysis was performed using Modified Intent-to-Treat method, defined as the proportions of participants meeting the response criteria in numerator and denominator based on all treated participants. The analysis was performed in all treated participants.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Part A: Peginterferon Lambda-1a + RBV + TVR (Open Label)
Number analyzed (Participants) | 27
Percentage of participants | 51.9 [31.9 to 71.3]

2. Primary Outcome: Percentage of Participants With Sustained Virologic Response at Follow-up Week 12 (SVR12) - Part B
Description: SVR12 was defined as Hepatitis C virus (HCV) RNA level below lower limit of quantitation, target detected or not detected at Week 12 of post-treatment follow-up. HCV RNA level was measured using the Roche COBAS® TaqMan HCV Test v.2.0 (lower limit of quantitation =25 IU/mL; limit of detection ~ 10 IU/mL).
Time Frame: Follow-up Week 12
Population: The analysis was performed using Modified Intent-to-Treat method defined as the proportions of participants meeting the response criteria in numerator and denominator based on all treated participants. The analysis was performed in all treated participants.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Part B: Peginterferon Lambda-1a + RBV + TVR | Part B: Peginterferon Alfa-2a + RBV + TVR
Number analyzed (Participants) | 411 | 206
Percentage of participants | 76.2 [72 to 80.3] | 82 [76.8 to 87.3]
Statistical Analysis 1: Comparison: Part B: Peginterferon Lambda-1a + RBV + TVR vs Part B: Peginterferon Alfa-2a + RBV + TVR; Test type: Non-Inferiority — Non-inferiority of Lambda/RBV/TVR to Alfa/RBV/TVR was not established because the lower limit of the 95% CI was less than the predefined non-inferiority margin of -12%. As a result, key secondary endpoints were not tested hierarchically to compare treatment groups; p = 0.0855, Mantel Haenszel — Non-inferiority testing is based on lower limit of confidence interval

3. Primary Outcome: Number of Participants With Adverse Events (AEs), Serious Adverse Events (SAEs), Drug Related AEs, Discontinuation Due to AEs, Dose Reductions and Death - Part A
Description: An AE was defined as any new untoward medical occurrence or worsening of a pre-existing medical condition in a participant or clinical investigation participant administered an investigational (medicinal product. An SAE was defined as any untoward medical occurrence that at any dose resulted in death, was life-threatening, required inpatient hospitalization or caused prolongation of existing hospitalization.
Time Frame: Day 1 of treatment up to Week 48
Population: Safety analysis included all treated participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Peginterferon Lambda-1a + RBV + TVR (Open Label)
Number analyzed (Participants) | 27
Participants
  AEs | 26
  SAEs | 6
  Drug related AEs | 12
  Discontinuation due to AEs | 2
  Death | 0
  Dose reductions - Lambda | 3
  Dose reductions - RBV | 7

4. Secondary Outcome: Percentage of Participants With Sustained Virologic Response at Follow-up Week 12 (SVR12) - Part A
Description: SVR12 was defined as Hepatitis C virus (HCV) RNA level below lower limit of quantitation (LLOQ), target detected or not detected at Week 12 of post-treatment follow-up. HCV RNA level was measured using the Roche COBAS® TaqMan HCV Test v.2.0 (LLOQ =25 IU/mL; limit of detection ~ 10 IU/mL).
Time Frame: Follow-up Week 12
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- Part A: Peginterferon Lambda-1a + RBV + TVR (Open Label): Participants were followed up for 48 weeks who received treatment as: Peginterferon Lambda-1a 180 mcg subcutaneously, once weekly for 24 or 48 weeks depending on the extended rapid virologic response (eRVR); Ribavirin 1000 or 1200 mg (based on weight) tablets, orally daily in 2 divided doses for 24 or 48 weeks depending on the eRVR response; Telaprevir 750 mg tablets, orally three times a day for 12 weeks.
Arm/Group | Part A: Peginterferon Lambda-1a + RBV + TVR (Open Label)
Number analyzed (Participants) | 27
Percentage of participants | 48.1 [28.7 to 68.1]

5. Secondary Outcome: Percentage of Subjects With Sustained Virologic Response at Follow-Up Week 24 (SVR24) - Part A
Description: SVR24 was defined as Hepatitis C virus (HCV) RNA level below lower limit of quantitation (LLOQ), target detected or not detected at Week 24 of post-treatment follow-up. HCV RNA level was measured using the Roche COBAS® TaqMan HCV Test v.2.0 (LLOQ) =25 IU/mL; limit of detection ~ 10 IU/mL). The analysis was performed using Modified Intent-to-Treat method defined as the proportions of participants meeting the response criteria in numerator and denominator based on all treated participants. The analysis was performed in all treated participants.
Time Frame: Follow up week 24
Population: Analysis was performed using Observed value method, defined as proportions of participants meeting response criteria in numerator and denominator - all treated participants with HCV RNA measured at follow-up Week 24. Analysis was performed in all treated participants with HCV RNA measured at follow-up Week 24 due to early study termination.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Part A: Peginterferon Lambda-1a + RBV + TVR (Open Label)
Number analyzed (Participants) | 27
Percentage of participants | 40.7 [22.4 to 61.2]

6. Secondary Outcome: Percentage of Treatment-Naïve Participants With Sustained Virologic Response at Follow-up Week 12 (SVR12) - Part B
Description: as for outcome 2
Time Frame: Follow-up Week 12
Population: The analysis was performed using Modified Intent-to-Treat method defined as the proportions of participants meeting the response criteria in numerator and denominator based on all treated participants. The analysis was performed in all treatment-naive treated participants.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Part B: Peginterferon Lambda-1a + RBV + TVR | Part B: Peginterferon Alfa-2a + RBV + TVR
Number analyzed (Participants) | 311 | 155
Percentage of participants | 73.6 [68.7 to 78.5] | 81.9 [75.9 to 88]

7. Secondary Outcome: Percentage of Participants With Treatment Emergent Cytopenic Abnormalities - Part B
Description: Cytopenic abnormalities included anemia defined as hemoglobin <10 grams/decilitre; neutropenia defined as Absolute neutrophil count (ANC) <750 cubic millimetre (mm^3); thrombocytopenia defined as platelets <50,000 mm^3.
Time Frame: After Day 1 of treatment up to Week 48
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Part B: Peginterferon Lambda-1a + RBV + TVR | Part B: Peginterferon Alfa-2a + RBV + TVR
Number analyzed (Participants) | 411 | 206
Percentage of participants | 11.7 [8.6 to 14.8] | 55.8 [49 to 62.6]

8. Secondary Outcome: Percentage of Participants With Extended Rapid Virologic Response (eRVR) - Part B
Description: as for outcome 1
Time Frame: Week 4 and Week 12
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Part B: Peginterferon Lambda-1a + RBV + TVR | Part B: Peginterferon Alfa-2a + RBV + TVR
Number analyzed (Participants) | 411 | 206
Percentage of participants | 64 [59.3 to 68.6] | 70.9 [64.7 to 77.1]

9. Secondary Outcome: Percentage of Participants With On-Treatment Flu-Like Symptoms And Musculoskeletal Symptoms- Part B
Description: Flu-like symptoms included pyrexia, chills, and pain. Musculoskeletal symptoms included arthralgia, myalgia, and back pain.
Time Frame: After Day 1 of treatment up to Week 48
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Part B: Peginterferon Lambda-1a + RBV + TVR | Part B: Peginterferon Alfa-2a + RBV + TVR
Number analyzed (Participants) | 411 | 206
Percentage of participants
  Flu-Like Symptoms | 14.4 [11 to 17.7] | 36.4 [29.8 to 43]
  Musculoskeletal symptoms | 21.4 [17.4 to 25.4] | 30.6 [24.3 to 36.9]

10. Secondary Outcome: Percentage of Participants With Sustained Virologic Response at Follow- upWeek 24 (SVR24) - Part B
Description: SVR24 was defined as Hepatitis C virus (HCV) RNA level below lower limit of quantitation (LLOQ), target detected or not detected at Week 24 of post-treatment follow-up. HCV RNA level was measured using the Roche COBAS® TaqMan HCV Test v.2.0 (LLOQ) =25 IU/mL; limit of detection ~ 10 IU/mL).
Time Frame: Follow-up Week 24
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Part B: Peginterferon Lambda-1a + RBV + TVR | Part B: Peginterferon Alfa-2a + RBV + TVR
Number analyzed (Participants) | 223 | 108
Percentage of participants | 83 [78 to 87.9] | 87 [80.7 to 93.4]

11. Secondary Outcome: Percentage of Participants With Rash
Description: All skin reactions involving rash or rash-like events that occurred on treatment were reported.
Time Frame: After Day 1 of treatment up to Week 48
Population: The analysis was performed in all treated participants.
Measure: Number; unit: Percentage of participants
Arm/Group | Part A: Peginterferon Lambda-1a + RBV + TVR (Open Label) | Part B: Peginterferon Lambda-1a + RBV + TVR | Part B: Peginterferon Alfa-2a + RBV + TVR
Number analyzed (Participants) | 27 | 411 | 206
Percentage of participants | 63 | 36.3 | 38.3

ADVERSE EVENTS:
Time Frame: Day 1 of treatment up to Week 48
Arm/Group | Part A: Peginterferon Lambda-1a + RBV + TVR (Open Label) | Part B: Peginterferon Lambda-1a + RBV + TVR | Part B: Peginterferon Alfa-2a + RBV + TVR
All-Cause Mortality (participants affected / at risk) | 0/27 | 1/411 | 1/206
Serious Adverse Events (participants affected / at risk) | 6/27 | 43/411 | 20/206
Other Adverse Events (participants affected / at risk) | 26/27 | 369/411 | 197/206
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part A: Peginterferon Lambda-1a + RBV + TVR (Open Label) (N=27) | Part B: Peginterferon Lambda-1a + RBV + TVR (N=411) | Part B: Peginterferon Alfa-2a + RBV + TVR (N=206)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Strangulated hernia (General disorders) | 0 (0) | 1 (1) | 0 (0)
Substance-induced psychotic disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Overdose (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Blood creatinine increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Electrocardiogram QT prolonged (Investigations) | 0 (0) | 1 (1) | 0 (0)
Hepatic enzyme increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Lipase increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Pancreatic enzymes increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Carotid bruit (Investigations) | 0 (0) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 3 (4)
Pancytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Demyelination (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Ocular icterus (Eye disorders) | 0 (0) | 3 (3) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Peptic ulcer haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 0 (0) | 2 (2) | 1 (1)
Ileus (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Gastrointestinal vascular malformation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Jaundice (Hepatobiliary disorders) | 3 (3) | 11 (11) | 2 (2)
Drug-induced liver injury (Hepatobiliary disorders) | 0 (0) | 4 (4) | 0 (0)
Hepatotoxicity (Hepatobiliary disorders) | 0 (0) | 2 (2) | 0 (0)
Hypertransaminasaemia (Hepatobiliary disorders) | 0 (0) | 2 (2) | 0 (0)
Jaundice cholestatic (Hepatobiliary disorders) | 0 (0) | 2 (2) | 0 (0)
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 5 (5)
Drug reaction with eosinophilia and systemic symptoms (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part A: Peginterferon Lambda-1a + RBV + TVR (Open Label) (N=27) | Part B: Peginterferon Lambda-1a + RBV + TVR (N=411) | Part B: Peginterferon Alfa-2a + RBV + TVR (N=206)
Amylase increased (Investigations) | 0 (0) | 21 (26) | 3 (5)
Blood bilirubin increased (Investigations) | 2 (3) | 19 (25) | 2 (2)
Alanine aminotransferase increased (Investigations) | 2 (2) | 30 (33) | 1 (2)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 30 (38) | 1 (2)
Bilirubin conjugated increased (Investigations) | 2 (2) | 6 (9) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 31 (34) | 37 (41)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 12 (13) | 24 (27)
Anaemia (Blood and lymphatic system disorders) | 3 (3) | 53 (55) | 100 (111)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 10 (17) | 35 (45)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 9 (13) | 32 (41)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (2) | 17 (22)
Headache (Nervous system disorders) | 8 (9) | 66 (76) | 42 (54)
Dizziness (Nervous system disorders) | 2 (2) | 52 (55) | 24 (33)
Dysgeusia (Nervous system disorders) | 3 (3) | 11 (11) | 9 (11)
Syncope (Nervous system disorders) | 2 (2) | 5 (5) | 1 (1)
Fatigue (General disorders) | 16 (16) | 143 (162) | 75 (92)
Asthenia (General disorders) | 0 (0) | 81 (95) | 61 (69)
Pyrexia (General disorders) | 2 (2) | 31 (37) | 53 (61)
Influenza like illness (General disorders) | 3 (4) | 26 (29) | 36 (39)
Chills (General disorders) | 1 (1) | 35 (42) | 35 (41)
Injection site reaction (General disorders) | 4 (4) | 7 (7) | 6 (6)
Pain (General disorders) | 2 (2) | 6 (6) | 6 (6)
Oedema peripheral (General disorders) | 2 (2) | 15 (16) | 3 (3)
Injection site rash (General disorders) | 3 (3) | 6 (6) | 0 (0)
Insomnia (Psychiatric disorders) | 8 (8) | 102 (110) | 56 (63)
Anxiety (Psychiatric disorders) | 0 (0) | 13 (14) | 11 (11)
Depression (Psychiatric disorders) | 5 (6) | 25 (26) | 11 (11)
Irritability (Psychiatric disorders) | 3 (3) | 33 (40) | 8 (8)
Nausea (Gastrointestinal disorders) | 11 (12) | 172 (195) | 67 (78)
Diarrhoea (Gastrointestinal disorders) | 13 (13) | 61 (70) | 37 (43)
Vomiting (Gastrointestinal disorders) | 5 (5) | 66 (93) | 25 (29)
Anal pruritus (Gastrointestinal disorders) | 4 (4) | 59 (64) | 22 (22)
Anorectal discomfort (Gastrointestinal disorders) | 5 (5) | 28 (30) | 17 (18)
Dyspepsia (Gastrointestinal disorders) | 2 (2) | 28 (30) | 13 (17)
Haemorrhoids (Gastrointestinal disorders) | 1 (1) | 17 (17) | 11 (11)
Proctalgia (Gastrointestinal disorders) | 2 (2) | 8 (9) | 5 (6)
Hyperbilirubinaemia (Hepatobiliary disorders) | 3 (3) | 44 (56) | 4 (4)
Pruritus (Skin and subcutaneous tissue disorders) | 13 (13) | 187 (209) | 100 (126)
Rash (Skin and subcutaneous tissue disorders) | 12 (13) | 123 (131) | 57 (62)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | 52 (56) | 27 (27)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1) | 9 (9) | 23 (24)
Rash generalised (Skin and subcutaneous tissue disorders) | 5 (5) | 4 (4) | 2 (2)
Skin exfoliation (Skin and subcutaneous tissue disorders) | 2 (2) | 4 (4) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 49 (58) | 43 (55)
Myalgia (Musculoskeletal and connective tissue disorders) | 4 (4) | 49 (61) | 43 (56)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 4 (4) | 14 (14) | 2 (2)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 85 (93) | 42 (47)
Hyperuricaemia (Metabolism and nutrition disorders) | 1 (1) | 32 (43) | 11 (11)
Upper respiratory tract infection (Infections and infestations) | 2 (2) | 3 (4) | 4 (4)
Gastroenteritis (Infections and infestations) | 2 (2) | 5 (5) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.